CLINICAL TRIAL: NCT02575495
Title: A Pilot Randomized Control Study of Shortening Antibiotic Treatment Duration For Asymptomatic Bacteriuria Within A Month After Kidney Transplantation
Brief Title: A Randomized Control Trial of Antibiotic Treatment Duration For Asymptomatic Bacteriuria After Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC_580278
Record Dates: First submitted 2015-10-08; First posted 2015-10-14 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Kidney Transplantation; Bacteriuria; Asymptomatic Infections
MeSH Terms: conditions — Bacteriuria; Asymptomatic Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7 days course of antibiotic treatment (Experimental): To assign the 7 days course of antibiotic treatment, start specific intravenous antibiotic therapy as microbiological susceptibility from urine culture
  Interventions: Drug: 7 days course of antibiotic treatment
- 14 days course of antibiotic treatment (Active Comparator): To assign the 14 days course of antibiotic treatment, start specific intravenous antibiotic therapy as microbiological susceptibility from urine culture
  Interventions: Drug: 14 days course of antibiotic treatment

INTERVENTIONS:
Drug: 7 days course of antibiotic treatment — start specific intravenous antibiotic therapy as microbiological susceptibility from urine culture for 7 days
  Other Names: short-course antibiotic treatment
  Arms: 7 days course of antibiotic treatment
Drug: 14 days course of antibiotic treatment — start specific intravenous antibiotic therapy as microbiological susceptibility from urine culture for 14 days
  Other Names: traditional-course antibiotic treatment
  Arms: 14 days course of antibiotic treatment

SUMMARY:
The major hypothesis to be tested is that there was no difference in the clinical outcome between 7(short-course) and 14(traditional-course) days of antibiotic treatment for asymptomatic bacteriuria early after kidney transplantation.

DETAILED DESCRIPTION:
Introduction: Treatment of asymptomatic bacteriuria is a common practice in renal transplant centers leading to prolong exposure of antimicrobial agents with long hospital length of stay. The duration of antibiotics treatment in this condition have never been proposed.

Objective: To evaluate the proper duration of antibiotic treatment for asymptomatic bacteriuria early (less than 1 month) after kidney transplantation

Method: This is a prospective, randomized, open labeled, single center study using intention to treat analysis. Patients will be identified and after informed consent is obtained, will be randomized to receive 7 or 14 days course of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* First kidney transplantation
* Asymptomatic bacteriuria

Exclusion Criteria:

* Refusal to participate in the study
* Re-transplantation or combined organ transplantation
* History of abnormal structure or function in native kidney, ureter and bladder system
* Kidney transplant recipients with history of recurrent urinary tract infection or incomplete course of urinary tract infection treatment before transplantation
* Hemodynamic unstable
* Urosepsis or other serious infectious complications(eg. symptomatic urinary tract infection/graft pyelonephritis, surgical site infection, infected urinoma/ hospital acquired pneumonia that mandates antibiotic therapy)
* Surgical complication (eg. anastomosis leakage, collection, ureteric stricture)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Composite end point of Symptomatic urinary tract infection, Sepsis, Graft function and Mortality rate | 1 month
  Composite end point at 1 month after discontinuing antibiotics

SECONDARY OUTCOMES:
Composite end point of Symptomatic urinary tract infection, Sepsis, Graft function and Mortality rate | 0.5 months
  Composite end point at 0.5 months after discontinuing antibiotics
Composite end point of Symptomatic urinary tract infection, Sepsis, Graft function and | 3 months
  Composite end point at 3 months after discontinuing antibiotics
duration of hospital stay | 30 days since randomization
  duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Pattraporn Ponglorpisit, MD, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Pattraporn Ponglorpisit, Ratchathewi, Bangkok, Thailand